CLINICAL TRIAL: NCT06833450
Title: Reliability of IUS in Crohn's Disease
Acronym: LOTUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0006
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease (CD)
Keywords: Crohn's disease; intestinal ultrasound; bowel wall thickness
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Transabdominal intestinal ultrasound — Transabdominal intestinal ultrasound

SUMMARY:
Transabdominal intestinal ultrasound (IUS) is gaining acceptance as a point-of-care test to objectively assess disease activity in Crohn's disease (CD).

In order to incorporate individual parameters in a future definition of transmural healing, and for the consistent application of IUS as a modality to assess treatment outcomes and establish therapeutic targets to ensure comparability between future studies, the inter-observer agreement should be determined for all relevant parameters.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease evolving for at least 1 months
* Patient older than 18 years
* Patient covered by French national health insurance
* Written informed consent

Exclusion Criteria:

* Pregnant women or breastfeeding
* Minor
* Patient deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of different IUS parameters between two operators | 1 year
  To assess in patients with CD the variability of IUS parameters between two operators

CONTACTS AND LOCATIONS:
Locations (1):
- CHU d'Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No